CLINICAL TRIAL: NCT00002219
Title: A Phase I/II, Open-Label, Multi-Center Study of the Pharmacokinetics, Safety, Tolerance and Activity of Two Dose Levels of Adefovir Dipivoxil (ADF) and Nelfinavir When Added to Antiretroviral Therapy for the Treatment of HIV-Infected Pediatric Patients
Brief Title: Safety and Effectiveness of Adding Adefovir Dipivoxil and Nelfinavir to the Anti-HIV Therapy of HIV-Infected Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 232H; GS-97-418
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-11

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Antiviral Agents; HIV Protease Inhibitors; Disease Progression; RNA, Viral; Adenine; Viral Load; Age Factors; Nelfinavir
MeSH Terms: conditions — HIV Infections; Disease Progression | interventions — Nelfinavir; Carnitine; adefovir dipivoxil

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Levocarnitine
Drug: Adefovir dipivoxil

SUMMARY:
The purpose of this study is to see if it is safe and effective to give adefovir (a new anti-HIV drug) plus nelfinavir to HIV-infected children who are already receiving other anti-HIV medications.

DETAILED DESCRIPTION:
During the first phase of the study (Days 1-6), the safety and tolerability of multiple doses of ADF is assessed when administered simultaneously with the patient's reverse transcriptase inhibitor (RTI) regimen. The second phase begins on Day 7 when nelfinavir is added to the therapy regimen for an additional 15 weeks. ADF pharmacokinetics are measured on Days 1, 2, and 7 (on a subset of 18 patients); peak and trough samples are collected on Day 28.

ELIGIBILITY:
Inclusion Criteria

Your child may be eligible for this study if he/she:

* Is 3 months to 16 years old.
* Is HIV-positive.
* Has never taken protease inhibitors or has previously taken ritonavir (RTV), saquinavir (SQV), or indinavir (IDV) and is willing to stop the medication at study entry.
* Is taking an anti-HIV drug combination that will not change during at least the 2 weeks prior to study entry.
* Agrees to use effective barrier methods of birth control, such as condoms, during the study.
* Has consent of parent or guardian.

Exclusion Criteria

Your child will not be eligible for this study if he/she:

* Has ever taken NFV.
* Has a history of opportunistic (AIDS-related) infection.
* Has any disease or illness that would prevent him/her from completing the study, including cancer.
* Has taken certain medications, including protease inhibitors at study entry.
* Is receiving an HIV vaccine at study entry.
* Is pregnant.

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - All Children's Hosp, St. Petersburg, Florida
  - Tulane Univ Med Ctr / Dept of Pediatrics, New Orleans, Louisiana
  - North Shore Univ Hosp / Division of Immunology, Great Neck, New York
  - St Lukes Roosevelt Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr / Dept of Pediatrics, The Bronx, New York
  - Duke Univ Med Ctr / Duke South Hosp, Durham, North Carolina
  - Med Univ of South Carolina, Charleston, South Carolina